CLINICAL TRIAL: NCT06513780
Title: A Study of the Correlation Between Portal Vein Thrombosis and Prognosis of Liver Transplantation
Status: Recruiting | Type: Observational
Sponsor: Ru-zhou Cai (Other)
Responsible Party: Sponsor-Investigator, Ru-zhou Cai, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: 2024-P2-187-01
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PVT: Participants who meet the inclusion criteria for portal vein thrombosis prior to liver transplantation
  Interventions: Other: Observation
- non-PVT: Participants who meet the inclusion criteria for the absence of portal vein thrombosis prior to liver transplantation.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention were made.

SUMMARY:
The goal of this observational study is to investigate the correlation between portal vein thrombosis (PVT) and the prognosis of liver transplantation. The main questions it aims to address are:

What is the prevalence of PVT? What are the risk factors associated with PVT? What is the prognostic impact of preoperative PVT on liver transplantation?

Participants are divided into two groups: the PVT group and the non-PVT group. The investigators will comparatively analyze the data of both groups, estimate the prevalence and risk factors of PVT, construct a predictive model for PVT that is applicable in clinical settings, and clarify the prognostic effects of PVT.

DETAILED DESCRIPTION:
The investigators aim to investigate the prevalence and risk factors of PVT, to develop a novel grading or rating system for PVT, and to explore the prognostic impact of preoperative PVT in liver transplantation.

The investigators will:

Recruit patients according to the inclusion/exclusion criteria and obtain signed informed consents. They will collect demographic and laboratory characteristics and classify patients into the PVT group and the non-PVT group based on preoperative ultrasound and/or computed tomography.

Collect patients' perioperative medical imaging, surgical procedures, pathology reports, postoperative treatments, follow-up data, and clinical endpoints.

Comparatively analyze the data of the PVT and non-PVT groups, estimate the prevalence and risk factors of PVT, construct a predictive model for PVT that is applicable in clinical settings, clarify the prognostic effects of PVT, and propose a grading/rating system for PVT.

ELIGIBILITY:
Inclusion Criteria:

1. Liver transplantation recipients
2. Aged 18 years or older.

Exclusion Criteria:

1. Retransplantation
2. Multi-organ transplantation
3. Portal vein tumor thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent in situ liver transplantation at the Liver Transplantation Center of Beijing Friendship Hospital affiliated with Capital Medical University from 2016-1-1 to 2025-12-31
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 10 years
  Rate of death from various causes after liver transplant
Postoperative portal vein thrombosis | 10 years
  Number of participants with portal vein thrombosis after liver transplant
Postoperative portal vein stenosis | 10 years
  Number of participants with portal vein stenosis after liver transplant

SECONDARY OUTCOMES:
Postoperative complications | 1 year
  Rate of re-surgery, interventional operation, endoscopy, dialysis, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No